CLINICAL TRIAL: NCT00214175
Title: Determination of Fraction Size Equivalent Dose (FED) Levels for Intracranial Conformal Avoidance Radiotherapy
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: RO04323; NCI-P01 CA88960
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Glioma; Brain Neoplasms
Keywords: low grade gliomas and benign CNS lesions
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients: patients who will receive XRT
- matched volunteers: Spouse or sibling

SUMMARY:
The primary objective is to evaluate and quantify the reproducibility of functional magnetic resonance imaging (fMRI) maps of the eloquent brain areas corresponding to specific neurological functions based on activation maps obtained with different thresholds in patients with benign and biopsy proven low-grade brain neoplasms. Another objective is to access the impairment in neurological function in image guided intracranial radiotherapy using neurocognitive assessment tools and to derive dose response curves relating the impairment in a particular neurological function to the FED received by the area of eloquent brain corresponding to it.

ELIGIBILITY:
Inclusion Criteria:

* Indication for brain radiotherapy.
* Ability to undergo MRI scans and time to participate in neurocognitive testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study patients will come from the population that is referred to radiotherapy for treatment of their low grade glioma or benign brain lesion and will undergo fractionated radiotherapy. The volunteers will be a spouse or sibling of a patient
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2004-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Tome, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States